CLINICAL TRIAL: NCT03609905
Title: A Phase I/II Randomized, Controlled, Clinical Trial for Assessment of the Safety and Efficacy of Allogeneic Adipose Mesenchymal Stem Cells in Moderate to Severe Ulcerative Colitis Patients
Brief Title: Adipose Mesenchymal Stem Cells (AMSC) for Treatment of Ulcerative Colitis
Acronym: AMSC_UC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liaocheng People's Hospital (Other)
Responsible Party: Principal Investigator, peng yan, Chief of gastroenterology, Liaocheng People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: lcsrmyy-yp1
Record Dates: First submitted 2018-06-01; First posted 2018-08-01 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Ulcerative Colitis (UC)
Keywords: ulcerative colitis (UC); mesenchymal stem cells(MSC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): interventions: The MSCs of 5×10*7 will be given in different sites within colonic submucosa at a total 100 ml with the use of the colonoscope. Once every week，a total of two times. Conventional drug therapy (5-amino-salicylic acid or glucocorticoid) is used
  Interventions: Biological: Adipose-cord mesenchymal stromal cells (A-MSCs); Other: Conventional drugs
- Control group (Other): interventions:Conventional drug therapy (5-amino-salicylic acid or glucocorticoid) is used
  Interventions: Other: Conventional drugs

INTERVENTIONS:
Biological: Adipose-cord mesenchymal stromal cells (A-MSCs) — A-MSCs 5 x 10~7 diluted on 100 mL of normal saline
  Arms: Intervention group
Other: Conventional drugs — 5-amino-salicylic acid or glucocorticoid

SUMMARY:
Ulcerative colitis is a form of inflammatory bowel disease characterized by diffuse inflammation of the colonic mucosa. It affects the rectum and extends proximally along a variable length of the colon. Ulcerative colitis is a chronic condition with a relapsing remitting course. Mesenchymal stem cells (MSCs) are a subset of adult stem cells residing in many tissues, including bone marrow (BM), adipose tissue, umbilical cord blood. Recent experimental findings have shown the ability of MSCs to home to damaged tissues and to produce paracrine factors with anti-inflammatory properties, potentially resulting in reduction of inflammation and functional recovery of the damaged tissues. The purpose of our study is to evaluate safety and efficacy of the intracolonic injection by using a colonoscope of allogeneic adipose MSCs in patients with moderate active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-65 years old
* Diagnosis of ulcerative colitis diagnosed at least 6 months earlier
* Moderate or severe activity defined by a Mayo score
* No serious infection, chronic diseases, diabetes and tuberculosis
* Unefficient by using 5-ASA, glucocorticoid or azathioprine
* Written informed consents were obtained from all subjects
* Capable of good communication with researchers and follow the entire test requirements
* Negative pregnancy test for women of childbearing potential (from menarche to menopause)

Exclusion Criteria:

* Pregnant or breastfeeding women or cognitively impaired adults
* History of malignant disease
* Infectious colitis
* Patients with known allergies to culture medium
* Patients having participated in clinical trials with any investigational drug within 1 month prior to enrolment in this study
* Patients with suspicion of Crohn's enterocolitis, indeterminate colitis, ischaemic colitis, radiation colitis, diverticular disease associated colitis, or microscopic colitis
* Patients with previous colectomy
* Positive to one or more of the infectious disease panel
* Treatment with surgery or biological treatment (infliximab or adamizumab) or Cyclosporine or tacrolimus or mycophenolate in the 8 weeks prior to inclusion in the study
* Presence of severe concomitant diseases
* Patients with clostridium difficult or cytomegalovirus infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Endoscopic Score (as Measured by Ulcerative Colitis Endoscopic Index of Severity) | Baseline, 8 weeks
  Ulcerative Colitis Endoscopic Index of Severity (UCEIS) is defined as Ulcerative Colitis Endoscopic Index of Severity, with higher scores indicating more severe disease

SECONDARY OUTCOMES:
Change from Baseline in clinical response (CDAI points) | Baseline, 8 weeks
  CDAI is defined as Clinical Disease Activity Index
To evaluate the quality of life index, Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | Baseline, 8 weeks
  The Short Inflammatory Bowel Disease Questionnaire (SIBDQ) is a health-related quality of life (HRQoL) tool measuring physical, social, and emotional status. It includes 10-item form of questions. Each question is scored on a Likert scale from 1 (worst) to 7 (best), scores from each item are summed to produce a total score, increased more than 3 scores were considered remission.
Histologic Evaluation of Ulcerative Colitis | Baseline, 8 weeks
  A 10 to 20 centimeter (cm) biopsy sample of inflamed mucosal tissue was taken from the worst affected area and scored using the Riley Index. The Riley Index is a histologic scoring system for the assessment of the activity and severity of ulcerative colitis, ranging from 0 to 24. It consists of 6 histologic features (acute inflammatory cell infiltrate, crypt abscesses, mucin depletion, surface epithelial integrity, chronic inflammatory cell infiltrate, and crypt architectural irregularities), all scored on a 4-point scale (higher scores indicate more severe disease).
Immune response in ulcerative colitis. | Baseline, 1, 4, 8 weeks
  A number of soluble mediators are detected, including proinflammatory cytokines (TNF, IFN-γ, IL-6.) and anti-inflammatory cytokines (IL-10, IL-4.).
Incidence of Treatment Adverse. | Baseline, 1, 4, 8 weeks
  An AE was any untoward medical occurrence in a participant

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yan, MD, Study Chair — Liaocheng People's Hospital
Locations (1):
- Liaocheng city people's hospital, Liaocheng, Shandong, China